CLINICAL TRIAL: NCT02486367
Title: Inflammation and Thrombosis in Patients With Severe Aortic Stenosis After Transcatheter Aortic Valve Replacement (TAVR)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Hospitals Cleveland Medical Center (Other)
Responsible Party: Principal Investigator, David A. Zidar, Assistant Professor of Medicine, University Hospitals Cleveland Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: UH IRB # 06-14-33
Record Dates: First submitted 2015-05-26; First posted 2015-07-01 (Estimated); Results first posted 2022-07-20 (Actual); Last update posted 2022-07-20 (Actual); Status verified 2022-06

CONDITIONS: Aortic Stenosis; Inflammation; Thrombosis
MeSH Terms: conditions — Aortic Valve Stenosis; Inflammation; Thrombosis | interventions — Clopidogrel; Ticagrelor

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Standard care/clopidogrel (Active Comparator): 300mg load followed by 75mg daily.
  Interventions: Drug: Clopidogrel
- Ticagrelor (Experimental): 180mg load followed by 90mg twice daily for 30 days.
  Interventions: Drug: Ticagrelor

INTERVENTIONS:
Drug: Clopidogrel — Standard ADP receptor blockade
  Arms: Standard care/clopidogrel
Drug: Ticagrelor — High potency ADP receptor blockade
  Arms: Ticagrelor

SUMMARY:
The central hypothesis of this study is that TAVR leads to platelet deposition and inflammatory cell activation that can be attenuated by the potent anti-platelet and/or pleiotropic effects of ticagrelor.

This single center, prospective randomized trial addresses the following specific aims:

1. To determine whether high-potency ADP receptor blockade reduces measures of platelet activation in patients after TAVR.
2. To determine whether high-potency ADP receptor blockade mitigates the pro-thrombotic inflammatory response observed after TAVR.

DETAILED DESCRIPTION:
BACKGROUND

Transcatheter Aortic Valve Replacement (TAVR) has emerged as an important alternative to surgical aortic valve replacement. While this technology represents an important advance over medical therapy or surgical AVR in poor operative candidates, the absolute mortality rates remain high, even in the great majority in whom an optimal hemodynamic result is achieved. In the randomized literature, the majority of these patients die within two years and two thirds of these deaths are due to cardiovascular (CV) events.

The mechanisms responsible for this limited survival are unclear from the clinical trials completed to date. While persistent valve disease undoubtedly plays a role in a subset of patients, particularly in patients with significant aortic regurgitation, the majority of events are due to non-valve related co-morbidities.

The hypothesis of this study is that TAVR results in at least three simultaneous CV insults: 1) the abrupt release of severely elevated left ventricular pressure into a non-compliant systemic vasculature leads to generalized endothelial cell activation, 2) the exposure of the pro-thrombotic and neo-antigenic contents of a degenerated aortic valve (known to histologically resemble atherosclerosis), and 3) the exposure of the replacement valve (bovine valve, stainless steel frame, polyester wrap). The investigators propose that these proximate events lead to platelet activation. Given the important link between thrombosis and inflammation governed by platelet-derived mediators and leukocyte-platelet interactions, they further hypothesize that monocyte activation is mediated, at least in part, by platelet-monocyte interactions, which has been shown to induce the expansion of inflammatory monocytes. Given the pro-thrombotic nature of inflammatory monocytes, they suspect a positive feedback loop may exist via the interplay of these thrombotic -inflammatory mechanisms, which may be abrogated via high potency ADP-receptor blockade.

TRIAL DESIGN Primary Objective of the Study This trial is designed to determine whether high-potency ADP-receptor blockade with ticagrelor, compared to standard care with clopidogrel, affects platelet responsiveness and the pattern of prothrombotic monocyte activation seen early after TAVR.

Primary and Secondary Outcomes The primary endpoint will be platelet responsiveness: platelet function will be measured one day after TAVR using the VerifyNow P2Y12 assay, and expressed in platelet reactivity units. The key secondary outcome measure will be the percentage of inflammatory monocytes, measured one day after TAVR. Inflammatory monocytes will be determined by flow cytometry, and expressed as a percentage of total monocytes.

ELIGIBILITY:
Inclusion Criteria:

1. Valvular heart disease and a clinical indication for TAVR
2. Age of 18 years or older
3. Capable of informed consent
4. Planned transfemoral TAVR

Exclusion Criteria:

1. Prior history of stroke, transient ischemic attack (TIA), or intracranial hemorrhage
2. Established bleeding diathesis or thrombocytopenia (<150k/dl)
3. End-stage renal disease
4. Severe hepatic impairment or liver cirrhosis
5. Pregnancy
6. Current infection
7. History of autoimmune disease
8. Established allergy to contrast agents, thienopyridines, aspirin, or ticagrelor
9. History of solid organ transplantation
10. Atrial Fibrillation, DVT, PE or other indication for long term anti-coagulation
11. Plan for direct aortic access or trans-apical TAVR
12. Enrollment in another clinical trial
13. Recent (< 12 months) or active excessive bleeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2015-06; Primary Completion 2019-01 (Actual); Study Completion 2019-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- UH Cleveland Medical Center, Cleveland, Ohio, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Standard Care/Clopidogrel | Ticagrelor
Started | 30 | 30
Completed | 30 | 30
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Standard Care/Clopidogrel | Ticagrelor | Total
Number analyzed (Participants) | 30 | 30 | 60
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 30 | 30 | 60
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 86 [80 to 90] | 85 [82 to 89] | 86 [82 to 90]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 20 | 34
  Male | 16 | 10 | 26
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 1 | 3
  White | 28 | 29 | 57
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Platelet Reactivity
Description: Platelet reactivity will be measured and reported as platelet reactivity units (PRU) using the VerifyNow system.
Time Frame: Day 0,1,7,&30
Population: Primary focus was Day 1. Day 7 and 30 were voluntary- not all participants came back.
Measure: Median (Standard Deviation); unit: Platelet Reactivity Units
Arm/Group | Standard Care/Clopidogrel | Ticagrelor
Number analyzed (Participants) | 30 | 30
Platelet Reactivity Units
  Day 0 | 275.5 (88.712) | 251 (78.725)
  Day 1 | 234 (80.956) | 128.5 (59.787)
  Day 7: number analyzed (Participants) | 27 | 26
  Day 7 | 208 (70.612) | 80 (89.424)
  Day 30: number analyzed (Participants) | 27 | 24
  Day 30 | 183 (60.044) | 134.5 (79.943)

2. Secondary Outcome: Inflammatory Monocyte Proportion
Description: The percentage of inflammatory (CD14+CD16+) monocytes as a proportion of total monocytes will be measured using flow cytometry on whole blood.
Time Frame: Day 0,1,7&30
Population: Primary focus was Day 1. Day 7 and 30 were voluntary- not all participants came back.
Measure: Median (Standard Deviation); unit: percentage of inflammatory monocyte
Arm/Group | Standard Care/Clopidogrel | Ticagrelor
Number analyzed (Participants) | 30 | 30
percentage of inflammatory monocyte
  Day 0 | 21.55103 (10.59286) | 21.50033 (10.45851)
  Day 1 | 22.23356 (9.344043) | 25.12275 (7.009391)
  Day 7: number analyzed (Participants) | 25 | 26
  Day 7 | 17.98342 (9.791872) | 21.626 (7.456207)
  Day 30: number analyzed (Participants) | 26 | 24
  Day 30 | 17.93496 (6.183553) | 21.06446 (7.326653)

3. Secondary Outcome: Change in D-Dimer Levels as Measured by Blood Test
Time Frame: Day 0,1,7,&30
Population: Primary focus was Day 1. Day 7 and 30 were voluntary- not all participants came back.
Measure: Median (Standard Deviation); unit: ng/mL
Arm/Group | Standard Care/Clopidogrel | Ticagrelor
Number analyzed (Participants) | 30 | 30
ng/mL
  Day 0 | 1564.668 (1070.615) | 1377.07 (129.768)
  Day 1: number analyzed (Participants) | 29 | 30
  Day 1 | 2851.912 (2024.33) | 2961.475 (2766.249)
  Day 7: number analyzed (Participants) | 27 | 26
  Day 7 | 2653.55 (1791.394) | 2635.958 (924.744)
  Day 30: number analyzed (Participants) | 26 | 22
  Day 30 | 1869.85 (1255.566) | 1554.43 (1641.397)

4. Secondary Outcome: Change in sCD14 as Measured by Blood Test.
Time Frame: Day 0,1,7,&30
Population: Primary focus was Day 1. Day 7 and 30 were voluntary- not all participants came back.
Measure: Median (Standard Deviation); unit: pg/mL
Arm/Group | Standard Care/Clopidogrel | Ticagrelor
Number analyzed (Participants) | 30 | 30
pg/mL
  Day 0 | 1638.721 (495.8533) | 1712.943 (515.0831)
  Day 1: number analyzed (Participants) | 29 | 30
  Day 1 | 1713.16 (657.8828) | 1896.489 (662.1276)
  Day 7: number analyzed (Participants) | 27 | 25
  Day 7 | 1765.934 (682.0759) | 1958.013 (734.3658)
  Day 30: number analyzed (Participants) | 26 | 22
  Day 30 | 1525.929 (527.5103) | 2077.568 (628.0957)

5. Secondary Outcome: Change in IL-6 as Measured by Blood Test.
Time Frame: Day 0,1,7,&30
Population: Primary focus was Day 1. Day 7 and 30 were voluntary- not all participants came back.
Measure: Median (Standard Deviation); unit: pg/mL
Arm/Group | Standard Care/Clopidogrel | Ticagrelor
Number analyzed (Participants) | 30 | 30
pg/mL
  Day 0 | 4.761 (7.661641) | 4.4 (7.997584)
  Day 1: number analyzed (Participants) | 29 | 30
  Day 1 | 43.127 (27.41416) | 52.125 (27.70069)
  Day 7: number analyzed (Participants) | 27 | 30
  Day 7 | 7.603 (49.1147) | 7.18502 (8.923163)
  Day 30: number analyzed (Participants) | 26 | 30
  Day 30 | 5.0825 (3.660653) | 4.511 (6.448078)

6. Secondary Outcome: Change in IL-8 as Measured by Blood Test
Time Frame: Day0,1,7,&30
Population: Primary focus was Day 1. Day 7 and 30 were voluntary- not all participants came back.
Measure: Median (Standard Deviation); unit: pg/mL
Arm/Group | Standard Care/Clopidogrel | Ticagrelor
Number analyzed (Participants) | 30 | 30
pg/mL
  Day 0 | 6.841063 (4.757768) | 4.837371 (5.069666)
  Day 1: number analyzed (Participants) | 29 | 30
  Day 1 | 8.58 (7.281141) | 7.558923 (12.75654)
  Day 7: number analyzed (Participants) | 27 | 26
  Day 7 | 4.98 (4.7204) | 4.584426 (5.476614)
  Day 30: number analyzed (Participants) | 26 | 22
  Day 30 | 4.81 (4.04262) | 3.783523 (6.472542)

7. Secondary Outcome: Change in Mono-CD62P as Measured by Blood Test
Time Frame: Day 0,1,7,&30
Population: Primary focus was Day 1. Day 7 and 30 were voluntary- not all participants came back.
Measure: Median (Standard Deviation); unit: percentage of monocytes
Arm/Group | Standard Care/Clopidogrel | Ticagrelor
Number analyzed (Participants) | 30 | 30
percentage of monocytes
  Day 0 | 1.675 (4.43711) | 1.525 (4.43853)
  Day 1 | 0.75 (2.47703) | 0.715 (1.82821)
  Day 7: number analyzed (Participants) | 25 | 26
  Day 7 | 0.69 (1.70967) | 0.73 (1.12174)
  Day 30: number analyzed (Participants) | 26 | 24
  Day 30 | 0.695 (0.4158) | 0.765 (0.70892)

8. Secondary Outcome: Change in Mono-2b3a as Measured by Blood Test
Time Frame: Day 0,1,7,&30
Population: Primary focus was Day 1. Day 7 and 30 were voluntary- not all participants came back.
Measure: Median (Standard Deviation); unit: percentage of monocytes
Arm/Group | Standard Care/Clopidogrel | Ticagrelor
Number analyzed (Participants) | 29 | 29
percentage of monocytes
  Day 0 | 2.27 (1.951142) | 1.45 (1.323815)
  Day 1 | 1.45 (2.310398) | 0.93 (1.215051)
  Day 7: number analyzed (Participants) | 26 | 25
  Day 7 | 0.615 (0.790469) | 1.23 (0.897987)
  Day 30: number analyzed (Participants) | 26 | 23
  Day 30 | 0.765 (2.268643) | 0.86 (1.522551)

ADVERSE EVENTS:
Time Frame: 30days
Arm/Group | Standard Care/Clopidogrel | Ticagrelor
All-Cause Mortality (participants affected / at risk) | 0/30 | 0/30
Serious Adverse Events (participants affected / at risk) | 11/30 | 8/30
Other Adverse Events (participants affected / at risk) | 0/30 | 0/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Standard Care/Clopidogrel (N=30) | Ticagrelor (N=30)
Major (TIMI3a or above) bleeding event (Blood and lymphatic system disorders) | 5 (5) | 5 (5)
Permanent pacemaker placement (Cardiac disorders) | 6 (6) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-01-31): https://cdn.clinicaltrials.gov/large-docs/67/NCT02486367/Prot_SAP_000.pdf